CLINICAL TRIAL: NCT03539939
Title: The Role of Smoking and Gingival Crevicular Fluid Markers on Coronally Advanced Flap Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: University of Louisville (Other)
Responsible Party: Principal Investigator, Nurcan Buduneli, Clinical Professor, Ege University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-DIS-004
Record Dates: First submitted 2018-05-15; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Gingival Recession; Smoking
Keywords: Gingival crevicular fluid; Gingival recession; Saliva; Smoking; Wound healing
MeSH Terms: conditions — Gingival Recession; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoker Group (Experimental): This group included smoker gingival recession patients.
  Interventions: Procedure: Coronally Advanced Flap
- Non-smoker Group (Active Comparator): This group included non-smoker gingival recession patients.
  Interventions: Procedure: Coronally Advanced Flap

INTERVENTIONS:
Procedure: Coronally Advanced Flap — The coronally advanced flap (CAF) is a procedure frequently used in periodontal plastic surgery. The main objective of this surgical technique is to mobilize the gingival margin and reposition it at a level more coronal (incisal direction) than its original location. CAF is mainly used for the treatment of gingival recessions.

SUMMARY:
Cigarette smoking is a patient-related factor that can affect healing of periodontal tissues and the success rate of root-coverage procedures. Neither the nature nor the mechanisms of action of cigarette smoking on root coverage are fully understood. Therefore, the hypothesis that cigarette smoking has negative impacts on the outcomes of root coverage after CAF surgery in systemically healthy individuals with an initial gingival thickness of at least 0.8 mm and who practice optimal oral hygiene was tested. It was also hypothesized that baseline analysis of disease-related biomarkers would shed light on the underlying mechanisms of a possible effect.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary central and lateral incisors, canines, and premolars and mandibular premolars with isolated buccal recessions classified as Miller Class I or II
* Study tooth should present tooth vitality, identifiable cemento-enamel junction (CEJ) and absence of caries, restorations or extensive non-carious cervical lesion.

Exclusion Criteria:

* Medical disorders such as diabetes mellitus, immunologic disorders, hepatitis
* History of previous mucogingival surgery at the gingival recession site
* Medications known to affect gingival tissues
* Antibiotic treatment in the past 6 months
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-05-03 (Actual); Primary Completion 2012-06-07 (Actual); Study Completion 2013-01-07 (Actual)

PRIMARY OUTCOMES:
Change in the percentage of root coverage | 1-month, 3-month and 6-month after coronally advanced flap (CAF)
  Root coverage were measured on digital photographs using specific software.

SECONDARY OUTCOMES:
Change in the percentage of complete root coverage | 1-month, 3-month and 6-month after coronally advanced flap (CAF)
Change in gingival thickness | Baseline,1-month, 3-month and 6-month after coronally advanced flap (CAF)
  Gingival thickness was measured with an ultrasonic device that uses the pulse echo principle. Ultrasonic pulses are transmitted at intervals of 1 millisecond through the sound-permeable mucosa and reflected, in part, at the surface of the alveolar bone or tooth attributable to different acoustic impedance. When an acoustic signal is transmitted within 2 to 3 seconds, gingival thickness is digitally displayed with a sensitivity of 0.01 mm.
Changing of the gingival crevicular fluid (GCF) biomarkers | Baseline,1-month, 3-month and 6-month after coronally advanced flap (CAF)
Changing of the salivary biomarkers | Baseline,1-month, 3-month and 6-month after coronally advanced flap (CAF)
Change in the visual analog scale (VAS) values | 1 to 7 day after coronally advanced flap (CAF)
  The visual analog scale (VAS) was used to evaluate pain during the postoperative follow-up period. It consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient selects a whole number (0-10 integers) that best reflects the intensity of their pain, with 0 being the no pain and 10 being the worst pain.